CLINICAL TRIAL: NCT06874166
Title: Social Cognition in Dystrophinopathies and Neurodevelopmental Disorders. Behavioural and Psychophisiological Measures
Brief Title: Social Cognition in Dystrophinopathies and Neurodevelopmental Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: L2-227
Record Dates: First submitted 2025-02-17; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Duchenne / Becker Muscular Dystrophy; Osteogenesis Imperfecta (OI); Social Cognition
Keywords: Social Cognition; Duchenne / Becker muscular dystrophy; Osteogenesis Imperfecta (OI); EEG; Interpersonal distance; Interoception
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Osteogenesis Imperfecta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- BMD/DMD group: Patients diagnosed with Duchenne and Becker muscular dystrophy (genetic and histological diagnosis and clinical diagnosis) (ambulant and non-ambulant), over the age of four.
  Interventions: Other: Electroencephalography (EEG); Other: Social Cognition Tasks
- OI group: Patients diagnosed with osteogenesis imperfecta, over the age of four.
  Interventions: Other: Electroencephalography (EEG); Other: Social Cognition Tasks
- Control group: Participants without any neurological or psychiatric disorder, over the age of four.
  Interventions: Other: Electroencephalography (EEG); Other: Social Cognition Tasks

INTERVENTIONS:
Other: Electroencephalography (EEG) — Recording of resting state EEG will be collected
Other: Social Cognition Tasks — Comfort-Distance Task: it will be used to measure the interpersonal comfort distance, the task will be implemented in immersive virtual reality environment Interoception will be measured through an auditory match task based on participants heart-beat A measure emotion processing will be collected through the emotion priming visual task, participants will be asked to detect trial by trial the target emotion which could be preceded by a congruent or incongruent visual priming

SUMMARY:
The primary aim of this observational study is to investigate specific aspects of social cognition in dystrophinopathies. Body awareness, interpersonal distance and emotional processing will be measured in a sample of patients affected by Becker (BMD) and Duchenne (DMD) muscular dystrophy, compared with a sample of patients affected by osteogenesis imperfecta (OI), and both compared with a control sample with typical development.

The secondary aim is to study cortical activity at rest, by means of electroencephalography (EEG), to explore frequencies and time course of EEG responses. Moreover, the relationship between EEG activity and neuropsychological, dispositional and subjective measures will be explored through correlational analyses.

DETAILED DESCRIPTION:
Study procedure includes: 1. Eligibility assessment according to inclusion and exclusion criteria. 2. Administration of questionnaires and scales for the characterization of cognitive and psychological features related with BMD/DMD and OI : Wechsler Intelligence Scale for Children 4th Edition (WISC-IV), Raven's Progressive Matrices; NEPSY-II; The Child Behavior Checklist (CBCL); PedsQL; Toronto Alexithymia Scale (TAS-20); Emotion Regulation Questionnaire (ERQ); Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA); Multidimensional Assessment of Interoceptive Awareness (MAIA); Body Shape Questionnaire (BSQ-14); and the Autism Spectrum Quotient (AQ, adult or child version) 3. Administration of experimental tasks. The Comfort-Distance Task (CDT) to measure the interpersonal comfort distance, the task will be implemented in immersive virtual reality by means of head-mounted displays (OCULUS ©2024 Meta). Interoceptive accuracy will be measured through a modified version of the heartbeat counting task. An emotional priming task will be administered in order to measure emotion processing, participants will be asked to detect trial by trial the target emotion which could be preceded by a congruent or incongruent visual priming.

All the tasks will be performed in a counterbalanced order, for an overall duration of about 40 minutes.

4. Recording of resting state EEG will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Duchenne and Becker muscular dystrophy (genetic and histological diagnosis and clinical diagnosis) (ambulant and non-ambulant).
* Patients diagnosed with osteogenesis imperfecta.
* Control group: participants without any neurological or psychiatric disorder

Exclusion Criteria:

* presence of comorbid diagnoses,
* sensory deficit
* specific condition that could prevent the application of the tests and tasks under study, such as: a) the need for PEG; b) the need for tracheostomy; c) the need for assisted ventilation.
* cognitive level lower than 60.

Min Age: 4 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For the statistical power analysis the size of the effect reported in Candini et al., 2017 (η2p = 0.28) has been considered, about the effect of diagnostic features on the peripersonal space, and the effect reported by Garcia et al., 2023 (η2p = 0.20) about the differences between DMD/BMD patients and neurotypicals in social cognition. The calculation, performed separately for the two different effects, returns a sample size between 17 and 23 minimum patients per group.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Interoception | Day 1
  interoceptive index
Interpersonal distance | Day 1
  Interpersonal comfort distance, measured in meters (m) within the virtual environment
Emotional processing | Day 1
  Visual priming task performance
EEG power | once
  EEG alpha power
EEG power | Day 1
  EEG beta power
EEG power | Day 1
  EEG theta power

IPD SHARING:
Plan to Share IPD: Undecided